CLINICAL TRIAL: NCT00005837
Title: Phase II Evaluation of Oxaliplatin in Persistent or Recurrent Squamous Cell Carcinoma of the Cervix
Brief Title: Oxaliplatin in Treating Patients With Recurrent or Refractory Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067852; GOG-127P
Record Dates: First submitted 2000-06-02; First posted 2003-05-05 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-07

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating patients who have recurrent or refractory cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of oxaliplatin by measuring response rate in patients with recurrent or refractory squamous cell carcinoma of the cervix who have failed on higher priority treatment protocols. II. Determine the nature and degree of toxicity of this drug in this patient population.

OUTLINE: Patients receive oxaliplatin IV over 2 hours. Treatment continues every 21 days for a maximum of 9 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed refractory or recurrent squamous cell carcinoma of the cervix that has failed local therapeutic measures and considered incurable Bidimensionally measurable disease Must not be eligible for a higher priority GOG protocol No known brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine normal Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: Not pregnant or nursing Fertile patients must use effective contraception No evidence of preexisting peripheral sensory neuropathy greater than CTC grade 1, including residual neuropathy attributed to prior chemotherapy and other chronic conditions (e.g., diabetes, venous stasis, and carpal tunnel syndrome) No history of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol directed chemotherapy No other uncontrolled concurrent illness (e.g., ongoing or active infection) No other malignancy within the past 5 years except nonmelanoma skin cancer and no other prior malignancy whose prior cancer treatment contraindicates this protocol therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony stimulating factors (CSFs) during first course of therapy At least 24 hours since prior CSFs during subsequent courses of therapy Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No prior oxaliplatin No more than 1 prior chemotherapy regimen Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: At least 3 weeks since prior surgery and recovered Other: At least 3 weeks since prior anticancer therapy and recovered No other concurrent investigational agents No concurrent antiretroviral therapy (HAART)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula M. Fracasso, MD, PhD, Study Chair — Washington University Siteman Cancer Center
Locations (72):
- United States (71):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Fracasso PM, Blessing JA, Wolf J, Rocereto TF, Berek JS, Waggoner S. Phase II evaluation of oxaliplatin in previously treated squamous cell carcinoma of the cervix: a gynecologic oncology group study. Gynecol Oncol. 2003 Jul;90(1):177-80. doi: 10.1016/s0090-8258(03)00253-1. PMID 12821360